CLINICAL TRIAL: NCT03827083
Title: Evaluation of Cognitive Functions by Cerebral Pulse Oximetry After General Anesthesia and Spinal Anesthesia in Geriatric Patients With Orthopedic Surgery
Brief Title: Evaluation of Cognitive Functions by Cerebral Pulse Oximetry
Status: Completed | Type: Observational
Sponsor: Tepecik Training and Research Hospital (Other)
Responsible Party: Principal Investigator, Fatih Mehmet Kurt, Principal İnvestigator, Tepecik Training and Research Hospital
Other Study IDs: Fatih Mehmet Kurt
Record Dates: First submitted 2019-01-04; First posted 2019-02-01 (Actual); Last update posted 2021-02-02 (Actual); Status verified 2021-02

CONDITIONS: Anesthesia; Cognitive Dysfunction
Keywords: spinal and general anesthesia; cerebral pulse oxymetry; cognitive dysfunction
MeSH Terms: conditions — Cognitive Dysfunction

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Spinal anesthesia: Evaluation of cognitive functions of patients under 65 years of age with lower extremity surgery by cerebral pulse oximetry
  Interventions: Other: cerebral pulse oximetry
- General anesthesia: Evaluation of cognitive functions of patients under 65 years of age with lower extremity surgery by cerebral pulse oximetry
  Interventions: Other: cerebral pulse oximetry

INTERVENTIONS:
Other: cerebral pulse oximetry — Cognitive Functions by Cerebral Pulse Oximetry After General Anesthesia and Spinal Anesthesia
  Other Names: postoperative cognitive dysfunctions

SUMMARY:
General and Spinal Anesthesia can be used in geriatric patients in orthopedic surgery. Post-op cognitive dysfunction can be seen in orthopedic surgeries in this group of patients.

In this study, the investigators aimed to compare cognitive functions between spinal and general anesthesia using cerebral and systemic oxygenation, hemodynamic data and pre-op, post-op cognitive function tests.

DETAILED DESCRIPTION:
Cerebral Oximeter is a monitoring application based on the measurement of regional oxygen saturation by transcutaneous route by near infrared spectroscopy technology. With this system that analyzes the intraparenchymal and microcirculation in the frontal cortex, cerebral oxygenation changes caused by possible hypoxemia are followed. Unlike pulse oximeter, it works in non-pulsatile conditions. In other words, continuous, real-time and safe oxygen saturation is continued to be measured even in the case of cardiopulmonary arrest. It is a significant advantage of noninvasive measurement according to jugular venous oxygen saturation measurement. For normal healthy people, the accepted normal range is 58-82%, while 0 to 15% of measurements are important for providing CPR process information.

Oxygen saturation measured by cerebral oximetry is different from that measured by other oxygen saturation measurement techniques. The main reason for this is the technique itself and the region where it is used. The radiation emitted by the cerebral oximetry sensor is aimed at the microvessel structure with venous and arterial mix. Since the contribution of venous and arterial blood volume in this structure is between 70-75% and 30-25%, different results are obtained based on only arterial or just venous bed measurements. In this sense, the measured saturation value is lower than the arterial oxygen and pulse oximetry saturation values; higher than venous values.

The ratio of oxyhemoglobin to the total hemoglobin below the region under evaluation of the system is expressed as, value in% System and reflected to the user as Regional Oxygen Saturation (rSO2). There are publications that can be used not only for cerebral but also for different tissues (ischemic limb, kidney, etc.).

General and Spinal Anesthesia can be used in geriatric patients in orthopedic surgery. Post-op cognitive dysfunction may be seen in orthopedic surgery in this patient group. There are not enough studies showing the correlation of cognitive functions with cerebral pulse oximetry after general and spinal anesthesia. In this study, the investigators aimed to compare cognitive functions between spinal and general anesthesia using cerebral and systemic oxygenation, hemodynamic data and pre-op, post-op cognitive function tests.

ELIGIBILITY:
Inclusion Criteria:

* ASA 1-2
* patients with lower extremity surgery
* Cognitive functions sufficient

Exclusion Criteria:

* Brain functions affected
* Peri-operative MAP <60 ones
* Those with electrolyte dysfunctions
* Those who need more blood and blood transfusion
* Patients with ASA 3 and above

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Study Population: Patients with lower extremity surgery, 65 years and older, ASA 1-2, Cognitive functions sufficient
Sampling Method: Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2019-01-09 (Actual); Primary Completion 2019-07-12 (Actual); Study Completion 2019-12-12 (Actual)

PRIMARY OUTCOMES:
mini-mental testing | preoperative and postoperative 48 hours mini-mental test change
  pre-op and post-op mini-mental testing
cerebral pulse oxymetry value | change in peroperative cerebral pulse oxymetry value
  peroperative cerebral pulse oxymetry value

SECONDARY OUTCOMES:
peripheral oxygen saturation | 1 min before induction, 1 min after induction or sedation, at surgical incision, 15 min of surgery, 30 min of surgery, 45 min of surgery, 60 min of surgery, leaving the operation room, at recovery and post-op 48 hours
  peripheral oxygen saturation
Heart rate | 1 min before induction, 1 min after induction or sedation, at surgical incision, 15 min of surgery, 30 min of surgery, 45 min of surgery, 60 min of surgery, leaving the operation room, at recovery and post-op 48 hours
  Heart rate
systolic blood pressure | 1 min before induction, 1 min after induction or sedation, at surgical incision, 15 min of surgery, 30 min of surgery, 45 min of surgery, 60 min of surgery, leaving the operation room, at recovery and post-op 48 hours
  systolic blood pressure
diastolic blood pressure | 1 min before induction, 1 min after induction or sedation, at surgical incision, 15 min of surgery, 30 min of surgery, 45 min of surgery, 60 min of surgery, leaving the operation room, at recovery and post-op 48 hours
  diastolic blood pressure
hemoglobin value | before 24 hours and after 24 hours of surgery
  hemoglobin value

CONTACTS AND LOCATIONS:
Overall Officials: Fatih Mehmet Kurt, MD, Principal Investigator — Tepecik Train and Research Hospital
Locations (1):
- İzmir Tepecik TRH, Izmir, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Papadopoulos G, Karanikolas M, Liarmakopoulou A, Papathanakos G, Korre M, Beris A. Cerebral oximetry and cognitive dysfunction in elderly patients undergoing surgery for hip fractures: a prospective observational study. Open Orthop J. 2012;6:400-5. doi: 10.2174/1874325001206010400. Epub 2012 Sep 3. PMID 22962570
- [Background] Guo JY, Fang JY, Xu SR, Wei M, Huang WQ. Effects of propofol versus sevoflurane on cerebral oxygenation and cognitive outcome in patients with impaired cerebral oxygenation. Ther Clin Risk Manag. 2016 Jan 18;12:81-5. doi: 10.2147/TCRM.S97066. eCollection 2016. PMID 26848269
- [Background] Kok WF, van Harten AE, Koene BM, Mariani MA, Koerts J, Tucha O, Absalom AR, Scheeren TW. A pilot study of cerebral tissue oxygenation and postoperative cognitive dysfunction among patients undergoing coronary artery bypass grafting randomised to surgery with or without cardiopulmonary bypass*. Anaesthesia. 2014 Jun;69(6):613-22. doi: 10.1111/anae.12634. Epub 2014 Apr 22. PMID 24750013
- [Background] Jo YY, Kim JY, Lee MG, Lee SG, Kwak HJ. Changes in cerebral oxygen saturation and early postoperative cognitive function after laparoscopic gastrectomy: a comparison with conventional open surgery. Korean J Anesthesiol. 2016 Feb;69(1):44-50. doi: 10.4097/kjae.2016.69.1.44. Epub 2016 Jan 28. PMID 26885301